CLINICAL TRIAL: NCT04526899
Title: Open-label, Randomized Phase II Trial With BNT111 and Cemiplimab in Combination or as Single Agents in Patients With Anti-PD-1-refractory/Relapsed, Unresectable Stage III or IV Melanoma
Brief Title: A Study to Investigate the Novel Agent BNT111 and Cemiplimab in Combination or as Single Agents in Patients With Advanced Melanoma That Has Not Responded to Other Forms of Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BNT111-01; 2020-002195-12 (EudraCT Number); 2023-509513-36-00 (EU CTIS Number)
Record Dates: First submitted 2020-08-18; First posted 2020-08-26 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Melanoma Stage III; Melanoma Stage IV; Unresectable Melanoma
Keywords: Cancer vaccine; Melanoma; Checkpoint inhibitor; Libtayo®; BNT111; Cemiplimab; RNA vaccine
MeSH Terms: conditions — Melanoma | interventions — cemiplimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BNT111 + cemiplimab (Experimental)
  Interventions: Biological: BNT111; Biological: Cemiplimab
- BNT111 monotherapy (Experimental)
  Interventions: Biological: BNT111
- Cemiplimab monotherapy (Experimental)
  Interventions: Biological: Cemiplimab

INTERVENTIONS:
Biological: BNT111 — IV injection
  Arms: BNT111 + cemiplimab; BNT111 monotherapy
Biological: Cemiplimab — IV infusion
  Arms: BNT111 + cemiplimab; Cemiplimab monotherapy

SUMMARY:
This is an open-label, randomized, multi-site, Phase II, interventional trial designed to evaluate the efficacy, tolerability, and safety of BNT111 + cemiplimab in anti-programmed death protein 1 (PD-1)/anti-programmed death ligand 1 (PD-L1)-refractory/relapsed patients with unresectable Stage III or IV melanoma. The contributions of BNT111 and cemiplimab will be delineated in single agent calibrator arms. Patients will be randomized in a 2:1:1 ratio to Arm 1 (BNT111 + cemiplimab) and calibrator Arm 2 (BNT111 monotherapy), and Arm 3 (cemiplimab monotherapy). Patients in single agent calibrator arms (Arms 2 and 3), who experience centrally verified disease progression under single agent treatment, may be offered addition of the other compound to the ongoing treatment after re-consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients must sign the written informed consent form (ICF) before any screening procedure.
* Patients must be aged >=18 years on the date of signing the informed consent.
* Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the trial.
* Patients must have histologically confirmed unresectable Stage III or IV (metastatic) cutaneous melanoma and measurable disease by RECIST v1.1.
* Patients must have confirmed disease progression on/after an approved anti-PD-1/PD-L1 regimen for melanoma as defined by RECIST v1.1.

  1. Previous exposure to approved anti-PD-1/PD-L1 containing regimen for at least 12 consecutive weeks and
  2. Current radiological progression to be confirmed by two scans 4 to 12 weeks apart. If progression is accompanied by new symptoms, or deterioration of performance status not attributed to toxicity, one scan is sufficient and
  3. Inclusion into this trial must be within 6 months of confirmation of disease progression on anti-PD-1/PD-L1 treatment, regardless of any intervening therapy.
* Patients should have received at least one but no more than five lines of prior therapy for advanced disease.
* Patients must be able to tolerate additional anti-PD-1/PD-L1 therapy (i.e., did not permanently discontinue anti-PD-1/PD-L1 therapy due to toxicity).
* Patients must have known B-Raf proto-oncogene (BRAF) mutation status.
* Patients with BRAF V600-positive tumor(s) should have received prior treatment with a BRAF inhibitor (alone or in combination with a mitogen-activated protein kinase kinase [MEK] inhibitor).

  * Note: Considering the possible negative impact of a prior BRAF/MEK therapy on immune system targeting therapies, patients with BRAF V600-positive tumors with no clinically significant tumor-related symptoms or evidence of rapid PD may be eligible for participation. This should be based on investigator assessment AND provided they are ineligible for, intolerant to, or have refused BRAF V600 mutation targeted therapy after receiving the information on possible other therapies including BRAF/MEK inhibitor-based therapy during the informed consent process.
* Patients must have an Eastern Cooperative Oncology Group performance status (PS) <=1.
* Adequate bone marrow function, as defined by hematological parameters (as defined in the protocol).
* Patients must have serum lactate dehydrogenase <= upper limit of normal.
* Patient should have adequate hepatic function, as defined in the protocol.
* Patient should have adequate kidney function, assessed by the estimated glomerular filtration rate >= 30 mL/min using the chronic kidney disease epidemiology collaboration equation.
* Patient should be stable with adequate coagulation, as defined in the protocol.
* Patients must provide the following biopsy samples:

  1. All patients: must provide a tumor tissue sample (formalin fixed paraffin-embedded [FFPE] blocks/slides) from a fresh biopsy collected before Visit Cycle1 Day1, or archival tissue. The archival tissue can be an FFPE block (not older than 3 years) or freshly cut slides (special storage conditions and immediate shipment to specialty lab are required), preferably derived from advanced disease stage.
  2. Patients at selected trial sites: After additional consent, patients must be amenable to pre-treatment and on-treatment peripheral blood mononuclear cell (PBMC) sampling and optional biopsy. If amenable, patients should provide a PBMC sample and optionally a biopsy which contains tumor tissue after failure/stop of last prior trial treatment.
* Women of childbearing potential (WOCBP) must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) at screening. Patients that are postmenopausal or permanently sterilized can be considered as not having reproductive potential. Female patients of reproductive potential must agree to use highly effective contraception during and for 6 months after the last trial drug administration.
* WOCBP must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during trial starting at screening, during the trial and for 6 months after receiving the last trial treatment.
* A man who is sexually active with a WOCBP and has not had a vasectomy must agree to use a barrier method of birth control, e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the trial and for 6 months after receiving the last trial treatment.

Exclusion Criteria:

* Patients must not be pregnant or breastfeeding.
* Patients must not have history of uveal, acral, or mucosal melanoma.
* Patients must have no ongoing or recent evidence (within the last 5 years) of significant autoimmune disease that required treatment with systemic immunosuppressive treatments which may pose a risk for irAEs.

  * Note: Patients with autoimmune-related hyperthyroidism, autoimmune-related hypothyroidism who are in remission, or on a stable dose of thyroid-replacement hormone, vitiligo, or psoriasis may be included.
* Patients must have no known primary immunodeficiencies, either cellular (e.g., DiGeorge syndrome, T cell-negative severe combined immunodeficiency [SCID]) or combined T and B cell immunodeficiencies (e.g., T and -B negative SCID, Wiskott Aldrich syndrome, ataxia telangiectasia, common variable immunodeficiency).
* Patients with uncontrolled type 1 diabetes mellitus or with uncontrolled adrenal insufficiency are not eligible.
* Patients must have no uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection; or diagnosis of immunodeficiency that is related to, or results in chronic infection. Mild cancer-related immunodeficiency (such as immunodeficiency treated with gamma globulin and without chronic or recurrent infection) is allowed.

  1. Patients with known HIV who have controlled infection (undetectable viral load and CD4 count above 350 either spontaneously or on a stable anti-viral regimen) are permitted. For patients with controlled HIV infection, monitoring will be performed per local standards.
  2. Patients with known hepatitis B virus (HBV) who have controlled infection (serum hepatitis B virus DNA polymerase chain reaction (PCR) that is below the limit of detection AND receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of HBV DNA per local standards. Patients must remain on anti-viral therapy for at least 6 months beyond the last dose of trial treatment.
  3. Patients who are known hepatitis C virus (HCV) antibody positive who have controlled infection (undetectable HCV RNA by PCR either spontaneously or in response to a successful prior course of anti-HCV therapy) are permitted.
  4. Patients with HIV or hepatitis must have their disease reviewed by the specialist (e.g., infectious disease specialist or hepatologist) managing this disease prior to commencing and throughout the duration of their participation in the trial.
* Patients with another primary malignancy that has not been in complete remission for at least 2 years, with the exception of those with a negligible risk of metastasis, progression or death (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, non-invasive, superficial bladder cancer or breast ductal carcinoma in situ).
* Current use or use within 3 months prior to trial enrollment of systemic immune suppression including:

  1. use of chronic systemic steroid medication (up to 5 mg/day prednisolone equivalent is allowed); patients using physiological replacement doses of prednisone for adrenal or pituitary insufficiency are eligible,
  2. other clinically relevant systemic immune suppression.
* Treatment with other anti-cancer therapy including chemotherapy, radiotherapy, investigational, or biological cancer therapy within 3 weeks prior to the first dose of trial treatment (6 weeks for nitrosureas). Adjuvant hormonotherapy used for breast cancer in long term remission is allowed.
* Current evidence of ongoing National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0) Grade > 1 toxicity of prior therapies before the start of treatment, with the exception of hair loss, hearing loss, Grade 2 peripheral neuropathy, or laboratory abnormalities not considered clinically significant per investigator's discretion, and those Grade 2 toxicities listed as permitted in other eligibility criteria.
* Patients who have a local infection (e.g., cellulitis, abscess) or systemic infection (e. g., pneumonia, septicemia) which requires systemic antibiotic treatment within 2 weeks prior to the first dose of trial treatment.
* Patients who have had a splenectomy.
* Patients who have had major surgery (e.g., requiring general anesthesia) within 4 weeks before screening, have not fully recovered from surgery, or have a surgery planned during the time of trial participation.
* Current evidence of new or growing brain or spinal metastases during screening. Patients with leptomeningeal disease are excluded. Patients with known brain or spinal metastases may be eligible if they:

  1. had radiotherapy or another appropriate therapy for the brain or spinal bone metastases,
  2. have no neurological symptoms that can be attributed to the current brain lesions,
  3. have stable brain or spinal disease on the computed tomography or magnetic resonance imaging scan within 4 weeks before randomization (confirmed by stable lesions on two scans at least 4 weeks apart, the second scan can be carried out during screening),
  4. do not require steroid therapy within 14 days before the first dose of trial treatment,
  5. spinal bone metastases are allowed, unless imminent fracture or cord compression is anticipated.
* History or current evidence of significant cardiovascular disease including, but not limited to:

  1. angina pectoris requiring anti-anginal medication, uncontrolled cardiac arrhythmia(s), severe conduction abnormality, or clinically significant valvular disease,
  2. QTc (F) prolongation > 480 ms,
  3. arterial thrombosis or pulmonary embolism within ≤ 6 months before the start of treatment,
  4. myocardial infarction within ≤ 6 months before the start of treatment,
  5. pericarditis (any NCI-CTCAE grade), pericardial effusion (NCI-CTCAE Grade >= 2), non-malignant pleural effusion (NCI-CTCAE Grade >=2) or malignant pleural effusion (NCI-CTCAE Grade >= 3) within <= 6 months before the start of treatment,
  6. Grade >= 3 symptomatic congestive heart failure (CHF) or New York Heart Association (NYHA) criteria Class >= II within <=6 months before the start of treatment.
* Patients who have received a live vaccine within 28 days of planned start of trial therapy.
* Known hypersensitivity to the active substances or to any of the excipients.
* Presence of a severe concurrent illness or other condition (e.g., psychological, family, sociological, or geographical circumstances) that does not permit adequate follow-up and compliance with the protocol.
* Prior treatment with BNT111 and/or with cemiplimab.

Inclusion criteria for entering add-on therapy

* Patients must have confirmed disease progression on monotherapy in Arm 2 or 3 of the trial.

  1. An initial radiological progression needs to be verified by BICR.
  2. Radiological progression to be confirmed by two scans 4 to 12 weeks apart unless initial progression is accompanied by new symptoms, or deterioration of PS not attributed to toxicity, in which case one scan is sufficient.
* Patients must sign a new ICF to continue with add-on therapy. Informed consent must be documented before any add-on-specific procedure is performed.
* WOCBP must have a negative serum (beta-hCG) at baseline. Patients that are postmenopausal or permanently sterilized can be considered as not having reproductive potential.
* Female patients of reproductive potential must agree to use adequate contraception during and for 6 months after the last trial drug administration.
* WOCBP must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during trial starting at screening, during the trial and for 6 months after receiving the last trial treatment.
* A man who is sexually active with a WOCBP and has not had a vasectomy must agree to use a barrier method of birth control, e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the trial and for 6 months after receiving the last trial treatment.

Exclusion criteria for entering add-on therapy

* Prior toxicity related to trial medication should have resolved to NCI-CTCAE v5.0 Grade ≤ 1 before the start of add-on treatment and may not have led to permanent discontinuation.
* The time between confirmed PD on monotherapy and start of add-on therapy shall not exceed 6 weeks.
* Current evidence of new or growing brain or spinal metastases at baseline (lesions that remained stable during initial treatment are allowed).
* Systemic immune suppression:

  1. use of chronic systemic steroid medication (up to 5 mg/day prednisolone equivalent is allowed); patients using physiological replacement doses of prednisone for adrenal or pituitary insufficiency are eligible,
  2. other clinically relevant systemic immune suppression.
* Presence of cardiovascular, renal, hepatic or any other disease that in the investigator's opinion, may increase the risks associated with trial participation or require treatments that may interfere with the conduct of the trial or the interpretation of trial results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2025-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (49):
- United States (6):
  - University Of Arizona College Of Medicine, Tucson, Arizona
  - University of California, San Francisco: Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Sylvester Comprehensive Cancer Center/ UMHC, Miami, Florida
  - Oncology Hematology West P.C. dba Nebraska Cancer Specialists, Omaha, Nebraska
  - Atlantic Health System / Morristown Medical Center, Morristown, New Jersey
  - Inova Dwight and Martha Schar Cancer Institute, Fairfax, Virginia
- Australia (3):
  - Border Medical Oncology, East Albury
  - Gold Coast Hospital, Southport
  - Melanoma Institute Australia, Sydney
- Germany (11):
  - Klinik für Dermatologie, Dermatochirurgie, Allergologie, Klinikum Bremen-Ost, Gesundheitnord GmbH, Bremen
  - Universitätsklinikum Essen (AoR), Essen
  - Universitätsklinikum Freiburg, Klinik füer Dermatologie und Venerologie, Freiburg im Breisgau
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Schleswig-Holstein (UKSH), Campus Kiel Hautkrebszentrum Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin der Johannes Gutenberg Universität Mainz KoeR, Mainz
  - Universitätsklinikum Mannheim GmbH, Mannheim
  - Klinikum Nürnberg Nord, Nuremberg
  - University Hospital Tübingen, Tübingen
  - Klinikum der Julius-Maximilians-Universität Würzburg, Würzburg
- Italy (9):
  - Istituto Di Ricovero E Cura A Carattere Scientifico - Istituto Tumori Giovanni Paolo Ii, Bari
  - Azienda ospedaliera universitaria Bologna, Bologna
  - Fondazione del Piemonte per l'Oncologia, Istituto di Candiolo (IRCCs), Candiolo
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumpori (IRST), Meldola
  - Istituto Nazionale Tumori Fondazione Pascale - IRCCS · S.C. Oncologia Medica Melanoma, Immunoterapia Oncologica e Terapie Innovative, Napoli
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua
  - Policlinico Universitario Campus Bio-Medico, Rome
  - Universita di Siena -Azienda Ospedaliera Universitaria Senese-Policlincio Santa Maria Alle Scotte, Siena
  - AOU Citta della Salute e della Scienza di Torino, Turin
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpital Specjalistyczny im. Luwika Rydygiera w Krakowie Sp. z o.o., Krakow
  - Zachodniopomorskie Centrum Onkologii, Szczecin
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Warsaw
- Spain (13):
  - Hospital Teresa Herrera (CHUAC), A Coruña
  - Hospital Universitari Germans Trias i Pujol (HUGTP), Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Institut Català d'Oncologia l'Hospitalet, Barcelona
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital General Universitario Gregorio Maranon, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Madrid
  - Hospital Universitario Marques De Valdecilla, Santander
  - Complejo Hospitalario Universitario De Santiago De Compostela, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Universitat de Valencia - Hospital Universitari i Politecnic La Fe de Valencia (Hospital La Fe Bulevar Sur), Valencia
- United Kingdom (3):
  - Beatson West of Scotland Cancer Centre - Greater Glasgow Health Board, Glasgow
  - The Christie - The Christie NHS Foundation Trust, Manchester
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total,184 participants were randomized to treatment but 3 participants (2 participants in Arm 1 and 1 participant in Arm 3, respectively) did not receive the study treatment.
Pre-assignment Details: Participants in Arms 2 and 3 who experienced centrally verified disease progression under single agent treatment were offered addition of the other compound to the ongoing treatment after re-consent. Participants of the two add-on treatment arms are a subset of the participants in Arm 2 and Arm 3, respectively.
Groups:
- Arm 1: BNT111 + Cemiplimab: Participants received BNT111 intravenous (IV) infusion once-weekly starting on Day 1 of Cycle 1 for the first 6 weeks, followed by once every 3 weeks (each cycle duration=21 days), along with Cemiplimab once every 3 weeks for up to 24 months or until confirmed progression of disease, withdrawal of consent or unacceptable toxicity, whichever occurs first.
- Arm 2: BNT111 Monotherapy: Participants received BNT111 IV infusion once-weekly starting on Day 1 of Cycle 1 for the first 6 weeks, followed by once every 3 weeks (each cycle duration=21 days), for up to 24 months or until confirmed progression of disease, withdrawal of consent or unacceptable toxicity, whichever occurs first. Participants in Arm 2 who experienced disease progression under monotherapy were eligible to continue with add-on therapy and received Cemiplimab once every 3 weeks as add-on treatment and BNT111 was continued according to the planned schedule. Participants received a total of 6 weekly injections during the initial trial treatment and the add-on therapy before moving to a once every 3-week schedule of injections.
- Arm 3: Cemiplimab Monotherapy: Participants received Cemiplimab IV infusion once every 3 weeks starting on Day 1 of Cycle 1 for up to 24 months or until confirmed progression of disease, withdrawal of consent or unacceptable toxicity, whichever occurs first. Participants in Arm 3 who experienced disease progression under monotherapy were eligible to continue with add-on therapy and received BNT111 once weekly for the first 6 weeks as add-on therapy, followed by treatments once every 3 weeks. Cemiplimab was given once every 3 weeks.
Period: Overall Study
Arm/Group | Arm 1: BNT111 + Cemiplimab | Arm 2: BNT111 Monotherapy | Arm 3: Cemiplimab Monotherapy
Started | 94 | 46 | 44
Treated | 92 | 46 | 43
Completed | 0 | 0 | 0
Not Completed | 94 | 46 | 44
Not completed — Withdrawal by Subject | 3 | 2 | 2
Not completed — Lost to Follow-up | 3 | 3 | 1
Not completed — Investigator's decision | 1 | 0 | 0
Not completed — Death | 33 | 17 | 13
Not completed — Other | 1 | 0 | 0
Not completed — On-Treatment | 19 | 10 | 12
Not completed — Survival Follow-up | 34 | 14 | 16

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent to treat (ITT) set that included all participants who were randomized.
Groups:
- Arm 1: BNT111 + Cemiplimab: Participants received BNT111 IV infusion once-weekly starting on Day 1 of Cycle 1 for the first 6 weeks, followed by once every 3 weeks (each cycle duration=21 days), along with Cemiplimab once every 3 weeks for up to 24 months or until confirmed progression of disease, withdrawal of consent or unacceptable toxicity, whichever occurs first.
- Arm 2: BNT111 Monotherapy: Participants received BNT111 IV infusion once-weekly starting on Day 1 of Cycle 1 for the first 6 weeks (each cycle duration=21 days), followed by once every 3 weeks for up to 24 months or until confirmed progression of disease, withdrawal of consent or unacceptable toxicity, whichever occurs first. Participants in Arm 2 who experienced disease progression under monotherapy were eligible to continue with add-on therapy and received Cemiplimab once every 3 weeks as add-on treatment and BNT111 was continued according to the planned schedule. Participants received a total of 6 weekly injections during the initial trial treatment and the add-on therapy before moving to a once every 3-week schedule of injections.
- Total: Total of all reporting groups
Arm/Group | Arm 1: BNT111 + Cemiplimab | Arm 2: BNT111 Monotherapy | Arm 3: Cemiplimab Monotherapy | Total
Number analyzed (Participants) | 94 | 46 | 44 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (13.54) | 63.1 (13.89) | 61.9 (15.78) | 62.7 (14.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 17 | 19 | 70
  Male | 60 | 29 | 25 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 7
  Not Hispanic or Latino | 85 | 41 | 41 | 167
  Unknown or Not Reported | 6 | 3 | 1 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 00 | 0
  White | 89 | 44 | 44 | 177
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Arm 1: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants in whom a complete response (CR) or partial response (PR) according to response evaluation criteria in solid tumors version 1.1 (RECIST v1.1) was observed as best overall response by blinded independent central review (BICR). Per RECIST 1.1 criteria, CR defined as the disappearance of all target lesions and PR was defined as the >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Up to 24 months
Population: Analysis was performed on modified intent to treat (mITT) set that included all participants who were randomized and had at least one dose of trial treatment and had a baseline and at least one post randomization tumor response assessment. Data for this outcome measure was planned for Arm 1 only and for other arms, results will be reported in secondary outcome measures after final analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: BNT111 + Cemiplimab
Number analyzed (Participants) | 89
percentage of participants | 18.0 [10.64 to 27.55]
Statistical Analysis 1: Comparison: Arm 1: BNT111 + Cemiplimab; Test type: Superiority; p = 0.0148, 1-sided exact binomial test

2. Secondary Outcome: Arms 2 & 3: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants in whom a CR or PR according to RECIST v1.1 observed as best overall response by BICR. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 24 Months
Reporting Status: Not Posted, anticipated posting 2026-12

3. Secondary Outcome: Duration of Response (DOR) As Assessed by Blinded Independent Central Review (BICR)
Description: DOR is defined as the time from first objective response (CR or PR) to first occurrence of objective tumor progression (progressive disease, PD) by BICR or death from any cause (whichever occurs first). Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 24 Months
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: Disease Control Rate (DCR) As Assessed by BICR
Description: DCR is defined as the percentage of participants in whom a CR, PR or stable disease (SD; assessed at least 6 weeks after first dose) is observed as best overall response by BICR. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 24 months
Reporting Status: Not Posted, anticipated posting 2026-12

5. Secondary Outcome: Time to Response (TTR) As Assessed by BICR
Description: TTR is defined as the time from randomization to the first objective tumor response (CR or PR) by BICR. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 24 months
Reporting Status: Not Posted, anticipated posting 2026-12

6. Secondary Outcome: Progression-Free Survival (PFS) As Assessed by BICR
Description: PFS is defined as the time from randomization to first objective tumor progression (PD) by BICR or death from any cause (whichever occurs first). Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 24 Months
Reporting Status: Not Posted, anticipated posting 2026-12

7. Secondary Outcome: Objective Response Rate (ORR) As Assessed by the Investigator
Description: ORR is defined as the percentage of participants in whom a CR or PR according to RECIST v1.1 observed as best overall response by investigator. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 24 months
Reporting Status: Not Posted, anticipated posting 2026-12

8. Secondary Outcome: Duration of Response (DOR) As Assessed by the Investigator
Description: as for outcome 3
Time Frame: Up to 24 Months
Reporting Status: Not Posted, anticipated posting 2026-12

9. Secondary Outcome: Disease Control Rate (DCR) As Assessed by the Investigator
Description: DCR defined as the percentage of participants in whom a CR, PR or stable disease (SD; assessed at least 6 weeks after first dose) is observed as best overall response by investigator. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 24 months
Reporting Status: Not Posted, anticipated posting 2026-12

10. Secondary Outcome: Time to Response (TTR) As Assessed by the Investigator
Description: TTR is defined as the time from randomization to the first objective tumor response (CR or PR) as assessed by investigator. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 24 months
Reporting Status: Not Posted, anticipated posting 2026-12

11. Secondary Outcome: Progression-Free Survival (PFS) As Assessed by the Investigator
Description: PFS is defined as the time from randomization to first objective tumor progression (PD) by investigator or death from any cause (whichever occurs first). Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 24 Months
Reporting Status: Not Posted, anticipated posting 2026-12

12. Secondary Outcome: Arm 1: Overall Survival (OS)
Description: OS is defined as the time from randomization to death from any cause. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 48 months
Reporting Status: Not Posted, anticipated posting 2026-12

13. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: A treatment-emergent adverse event (TEAE) is defined as any AE with an onset date on or after the first administration of trial treatment (if the AE was absent before the first administration of trial treatment) or worsened after the first administration of trial treatment (if the AE was present before the first administration of trial treatment). Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 27 months
Reporting Status: Not Posted, anticipated posting 2026-12

14. Secondary Outcome: Number of Participants With Immune-Related Adverse Events (irAE)
Description: AEs related to the use of immune checkpoint inhibitor (ICI) therapy are defined as immune-related (IR) AEs (irAEs). Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 27 months
Reporting Status: Not Posted, anticipated posting 2026-12

15. Secondary Outcome: Number of Participants Reporting Dose Reduction and Discontinuation Due to TEAE
Description: Participants with dose reduction and discontinuation due to TEAE will be reported. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 27 months
Reporting Status: Not Posted, anticipated posting 2026-12

16. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Hematology: Basophils
Description: Blood samples will be collected for the assessment of hematology parameters. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

17. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Hematology: Eosinophils
Description: as for outcome 16
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

18. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Hematocrit
Description: as for outcome 16
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

19. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Hemoglobin
Description: as for outcome 16
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

20. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Hematology: Lymphocytes
Description: as for outcome 16
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

21. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Clinical Chemistry: Albumin
Description: Blood samples will be collected for the assessment of clinical chemistry parameters. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

22. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Clinical Chemistry: Alkaline Phosphatase
Description: as for outcome 21
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

23. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Clinical Chemistry: Alanine Aminotransferase
Description: as for outcome 21
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

24. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Clinical Chemistry: Amylase
Description: as for outcome 21
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

25. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Clinical Chemistry: Aspartate Aminotransferase
Description: as for outcome 21
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

26. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Clinical Chemistry: Bilirubin
Description: as for outcome 21
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

27. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Clinical Chemistry: Creatine Kinase
Description: as for outcome 21
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

28. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Clinical Chemistry: Creatinine
Description: as for outcome 21
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

29. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Clinical Chemistry: C-Reactive Protein
Description: as for outcome 21
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

30. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Coagulation Factors: Activated Partial Thromboplastin Time
Description: Blood samples will be collected for the assessment of coagulation factors. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

31. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Coagulation Factors: Prothrombin Time
Description: as for outcome 30
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

32. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Endocrine Tests: Thyroxine
Description: Blood samples will be collected for the assessment of endocrine tests. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

33. Secondary Outcome: Change From Baseline in Laboratory Parameters Values: Urinalysis: pH
Description: Urine samples will be collected for the assessment of pH. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

34. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Parameters
Description: Participants with clinically significant abnormalities in laboratory parameters will be reported. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

35. Secondary Outcome: Change From Baseline in Vital Signs Parameters: Systolic Blood Pressure
Description: Systolic blood pressure (in mmHg) will be assessed. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

36. Secondary Outcome: Change From Baseline in Vital Signs Parameters: Diastolic Blood Pressure
Description: Diastolic blood pressure (in mmHg) will be assessed. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

37. Secondary Outcome: Change From Baseline in Vital Signs Parameters: Heart Rate
Description: Heart rate (in beats per minute) will be assessed. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

38. Secondary Outcome: Change From Baseline in Vital Signs Parameters: Respiratory Rate
Description: Respiratory Rate (in breaths per minute) will be assessed. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

39. Secondary Outcome: Change From Baseline in Vital Signs Parameters: Body Temperature
Description: Body Temperature (in degree Celsius) will be assessed. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

40. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Vital Signs
Description: Participants with clinically significant abnormalities in vital sign parameters will be reported. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

41. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 Items (EORTC QLQ-C30) Global Health Status Total Score
Description: Mean change from baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 Items (EORTC QLQ-C30) Global Health Status Score will be reported. Each item, except Global Health Status, is answered on a four-point scale (1-4): 1-not at all, 2-a little, 3-quite a bit, 4-very much. Response to Global Health Status is measured on a 1 to 7 scale. "1" being very poor and "7" being excellent. Positive changes indicated better health status or functioning, and negative changes indicated worsening of health status or functioning. Scale scores range from 0 to 100. Raw data was linearly transformed to be in a range from 0-100 where a higher score represents good health status, while lower scores indicate poor health status. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

42. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Functional Scales Score
Description: The EORTC QLQ-C30 questionnaire incorporates nine multi-item scales: 5 functional scales (physical, cognitive, role, emotional, and social); 3 symptom scales (pain, fatigue, and appetite loss) and a Global Health Status/QoL scale. EORTC QLQ-C30 Physical Functioning Score is a questionnaire to assess quality of life of cancer patients. It is composed of 30 items, multi-item measure (28 items) and 2 single-item measures. For the multiple item measure, 4-point scale is used and the score for each item range from "1 = not at all" to "4 = very much". Higher scores indicate worsening of symptoms. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

43. Secondary Outcome: Changes From Baseline in EORTC QLQ-C30 Symptoms Scales Score
Description: The EORTC QLQ-C30 questionnaire incorporates nine multi-item scales: 5 functional scales (physical, cognitive, role, emotional, and social); 3 symptom scales (pain, fatigue, and appetite loss) and a Global Health Status/QoL scale. Each item, except Global Health Status, is answered on a four-point scale (1-4): 1-not at all, 2-a little, 3-quite a bit, 4-very much. Each scale (symptom scale [pain, fatigue, and appetite loss] and Global Health Status/Quality of Life [QoL] scale) was linearly transformed to be in range from 0-100 where a higher score represents good health status, while lower scores indicate poor health status. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: From Baseline up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

44. Secondary Outcome: Time to First Clinically Meaningful Deterioration in Global Health Status Score as Measured by EORTC QLQ-C30
Description: Time to first clinically meaningful deterioration in global health status score as measured by EORTC QLQ-C30 will be reported. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

45. Secondary Outcome: Time to First Clinically Meaningful Deterioration in Symptoms and Functioning as Measured by EORTC QLQ-C30
Description: Time to first clinically meaningful deterioration in symptoms and functioning as measured by EORTC QLQ-C30 will be reported. Data for this outcome measure will be reported at the time of final results posting.
Time Frame: Up to 25 months
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: From Baseline until last dose of study treatment (up to 25 months). As per protocol, non-serious adverse events (AEs) with an onset date more than 90 days after last administration of study treatment are only reported below if assessed as related to investigational medicinal product by investigator.
Description: All-cause mortality analysis was performed on all randomized participants. One participant in Arm 3 died before treatment was started.
  As per protocol, analysis of serious AEs and other AEs was performed on the safety set, i.e., all participants who received study treatment (i.e., at least one dose of BNT111 or cemiplimab).
  Events that occurred in participants after add-on treatment was started, are presented in respective add-on treatment arms to avoid duplication of data.
Groups:
- Arm 2: BNT111 Monotherapy: Participants received BNT111 IV infusion once-weekly starting on Day 1 of Cycle 1 for the first 6 weeks, followed by once every 3 weeks (each cycle duration=21 days), for up to 24 months or until confirmed progression of disease, withdrawal of consent or unacceptable toxicity, whichever occurs first. Safety data included in this reporting group is until start of the add-on treatment.
- Arm 3: Cemiplimab Monotherapy: Participants received Cemiplimab IV infusion once every 3 weeks starting on Day 1 of Cycle 1 for up to 24 months or until confirmed progression of disease, withdrawal of consent or unacceptable toxicity, whichever occurs first. Safety data included in this reporting group is until start of the add-on treatment.
- Add-on Treatment: BNT111 + Cemiplimab (add-on): Participants in Arm 2 who experienced disease progression under monotherapy were eligible to continue with add-on therapy and received Cemiplimab once every 3 weeks as add-on treatment and BNT111 was continued according to the planned schedule. Participants received a total of 6 weekly injections during the initial trial treatment and the add-on therapy before moving to a once every 3-week schedule of injections. Participants included are a subset of Arm 2. Safety data included in this reporting group is from start of the add-on treatment until end of data collection.
- Add-on Treatment: Cemiplimab + BNT111 (add-on): Participants in Arm 3 who experienced disease progression under monotherapy were eligible to continue with add-on therapy and received BNT111 once weekly for the first 6 weeks as add-on therapy, followed by treatments once every 3 weeks. Cemiplimab was given once every 3 weeks. Participants included are a subset of Arm 3. Safety data included in this reporting group is from start of the add-on treatment until end of data collection.
Arm/Group | Arm 1: BNT111 + Cemiplimab | Arm 2: BNT111 Monotherapy | Arm 3: Cemiplimab Monotherapy | Add-on Treatment: BNT111 + Cemiplimab (add-on) | Add-on Treatment: Cemiplimab + BNT111 (add-on)
All-Cause Mortality (participants affected / at risk) | 33/94 | 6/46 | 6/44 | 11/25 | 7/22
Serious Adverse Events (participants affected / at risk) | 30/92 | 8/46 | 11/43 | 6/25 | 7/22
Other Adverse Events (participants affected / at risk) | 89/92 | 43/46 | 33/43 | 22/25 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: BNT111 + Cemiplimab (N=92) | Arm 2: BNT111 Monotherapy (N=46) | Arm 3: Cemiplimab Monotherapy (N=43) | Add-on Treatment: BNT111 + Cemiplimab (add-on) (N=25) | Add-on Treatment: Cemiplimab + BNT111 (add-on) (N=22)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 0 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0 | 0 | 0 | 0
Immune-mediated adrenal insufficiency (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Amaurosis fugax (Eye disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 8 | 1 | 3 | 3 | 2
Drug withdrawal syndrome (General disorders) | 0 | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 2 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 0 | 0 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Immune-mediated hepatitis (Hepatobiliary disorders) | 2 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 5 | 0 | 0 | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Bursa injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 1 | 0 | 0 | 0 | 0
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: BNT111 + Cemiplimab (N=92) | Arm 2: BNT111 Monotherapy (N=46) | Arm 3: Cemiplimab Monotherapy (N=43) | Add-on Treatment: BNT111 + Cemiplimab (add-on) (N=25) | Add-on Treatment: Cemiplimab + BNT111 (add-on) (N=22)
Anaemia (Blood and lymphatic system disorders) | 11 | 4 | 5 | 2 | 4
Sinus tachycardia (Cardiac disorders) | 5 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 2 | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 7 | 3 | 2 | 2 | 1
Constipation (Gastrointestinal disorders) | 9 | 2 | 4 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 7 | 7 | 4 | 3 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 34 | 11 | 6 | 3 | 5
Vomiting (Gastrointestinal disorders) | 23 | 6 | 5 | 3 | 4
Asthenia (General disorders) | 13 | 7 | 6 | 8 | 7
Axillary pain (General disorders) | 0 | 1 | 0 | 2 | 0
Chills (General disorders) | 45 | 24 | 2 | 5 | 14
Fatigue (General disorders) | 22 | 7 | 2 | 5 | 2
Influenza like illness (General disorders) | 20 | 10 | 0 | 2 | 1
Pyrexia (General disorders) | 66 | 35 | 2 | 12 | 17
Temperature regulation disorder (General disorders) | 1 | 2 | 0 | 2 | 1
Cytokine release syndrome (Immune system disorders) | 5 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 5 | 4 | 4 | 1 | 2
Oral herpes (Infections and infestations) | 3 | 4 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 5 | 2 | 2 | 3 | 1
Amylase increased (Investigations) | 2 | 3 | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 4 | 1 | 1 | 2
Blood alkaline phosphatase increased (Investigations) | 5 | 1 | 1 | 2 | 0
Blood chloride increased (Investigations) | 0 | 2 | 3 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 3 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 3 | 4 | 2 | 3
Blood magnesium decreased (Investigations) | 0 | 1 | 1 | 0 | 2
Blood phosphorus increased (Investigations) | 0 | 0 | 3 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 1 | 2 | 0 | 3
C-reactive protein increased (Investigations) | 1 | 1 | 6 | 2 | 4
Gamma-glutamyltransferase increased (Investigations) | 2 | 3 | 1 | 0 | 1
Lipase increased (Investigations) | 8 | 1 | 3 | 1 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 4 | 1 | 2
Platelet count increased (Investigations) | 0 | 0 | 2 | 0 | 2
Transaminases increased (Investigations) | 0 | 1 | 0 | 2 | 1
Weight decreased (Investigations) | 7 | 1 | 2 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 5 | 4 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 8 | 3 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 3 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 3 | 2 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 6 | 2 | 2 | 1
Dizziness (Nervous system disorders) | 6 | 3 | 2 | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 0 | 3 | 0 | 0
Headache (Nervous system disorders) | 11 | 6 | 1 | 1 | 2
Insomnia (Psychiatric disorders) | 4 | 1 | 4 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 5 | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 2 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 2 | 3 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 9 | 1 | 1 | 1 | 1
Hypertension (Vascular disorders) | 8 | 4 | 3 | 3 | 0
Hypotension (Vascular disorders) | 9 | 8 | 1 | 0 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this trial may be published or presented at scientific meetings. If this is foreseen, the investigator agrees to submit all manuscripts or abstracts to the sponsor before submission. This allows the sponsor to protect proprietary information and to provide comments. The sponsor will comply with the requirements for publication of trial results.

DOCUMENTS (2):
  • Study Protocol (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT04526899/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT04526899/SAP_001.pdf